CLINICAL TRIAL: NCT04570605
Title: Feasibility of Home Parasacral Transcutaneous Electrical Nerve Stimulation (PTENS) for the Voiding Dysfunction in the Pediatric Population: A Pilot Study
Brief Title: Feasibility of Parasacral Transcutaneous Electrical Nerve Stimulation PTENS for Voiding Dysfunction in Peds Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Glen Lau, Assistant Professor of Surgery, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 117756
Record Dates: First submitted 2019-04-19; First posted 2020-09-30 (Actual); Results first posted 2022-03-08 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Overactive Bladder; Voiding Disorders; Incontinence, Urinary
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Masking Description: patients will be randomized to standard urotherapy or urotherapy + PTENS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard Urotherapy (Active Comparator): Patients who meet eligibility criteria who will be counselled on standard recommendations for bladder management.
  Interventions: Other: Standard Urotherapy
- Standard Urotherapy + PTENS (Experimental): Patients who meet eligibility criteria who will be counselled on standard recommendations for bladder management AND use parasacral percutaneous TENS as additional treatment.
  Interventions: Device: parasacral transcutaneous electrical nerve stimulation (PTENS); Other: Standard Urotherapy

INTERVENTIONS:
Device: parasacral transcutaneous electrical nerve stimulation (PTENS) — electrode patches placed on skin of lower back just above each side of the gluteal cleft (parasacral) and attached to TENS unit at specific settings three times a week for 30 minutes for 12 weeks.
  Arms: Standard Urotherapy + PTENS
Other: Standard Urotherapy — standard behavioral therapy recommendations including timed voiding, fluid intake recommendations and bowel management recommendations including videos instructing patients and parents on these issues. This is current standard of care.

SUMMARY:
Pilot study for determining feasibility of home parasacral transcutaneous electrical nerve stimulation in treatment of urinary urgency and incontinence.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is the most common voiding dysfunction in children1. While many children may outgrow these issues, for some these symptoms persists and can lead to emotional, social, behavioral and physical problems. Multiple treatments exist for OAB but rarely is there guaranteed success. Many behavioral and lifestyle treatments involve a significant time investment and office visits on the part of the patient and family. Furthermore, medication therapy is often associated with bothersome side effects and is discontinued, even despite efficacy2. As such, treatments with potentially less adverse effects, often used in adult urology, are making their way into the pediatric urology practice. These include intravesical botulinum toxin injections, sacral nerve stimulation (SNS) and percutaneous tibial nerve stimulation (PTNS).

PTNS, first cleared by the United States Food and Drug Administration (FDA) in 2011 for adult use, has evolved into transcutaneous nerve stimulation in the pediatric population; obviating the need for needles during treatment. Studies suggest mixed efficacy in electric nerve stimulation for overactive bladder in the pediatric population, owing largely to the marked heterogeneity in treatment protocols. While some researchers follow the traditional tibial nerve pathway, others take a cue from SNS and target the parasacral area, while still others rely on signaling from even further peripheral nerves to modulate bladder overactivity 3-5. Perhaps further contributing to the disparate data is the varying treatment schedules used. Some centers perform treatments daily, others weekly, others twice or thrice a week. Similarly, some physicians recommend twenty-minute treatments, while others thirty or even sixty minutes. The majority of studies rely on an office-based treatment model, while a few have explored in home treatments 3-5. In the United States, there has been no study examining the feasibility or efficacy of home parasacral transcutaneous electric nerve stimulation (PTENS) on pediatric voiding dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Toilet trained (age 6) to age 17
* Diagnosis of urinary dysfunction, voiding dysfunction, overactive bladder, urgency incontinence, nocturnal enuresis. (These patients may also have an element of bowel dysfunction; however, we will not include a patient who had ONLY bowel dysfunction and NOT a voiding dysfunction).

Exclusion Criteria:

* Known neurologic diagnosis - such as myelomeningocele, caudal regression
* Known seizure disorder
* Age < 6 or > 17
* Lack of follow-up within 6 months of treatment
* Pacemaker, vagal nerve stimulator, or other implanted electrical device
* Intolerance of electrical nerve stimulation
* Pregnancy
* Implanted metal hardware
* Open sores or wounds over the sacral area
* Currently catheterizing for bladder drainage
* Known anatomic lower urinary tract abnormality (may be congenital or iatrogenic)
* Bowel only voiding dysfunction (Constipation ICD-10 K59.00)
* Non-English speaking families
* Families with health literacy precluding completion of questionnaires and voiding diaries
* Concurrent use of anticholinergics, alpha blockers or beta agonists for urologic treatments
* Untreated urinary tract infection

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glen A Lau, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah/Primary Children's Pediatric Urology, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be stored on password protected computers in the facility and collected data will be entered in a REDCap database. Individual participant data will not be shared with any individuals other than the study personnel as only these individuals will have access to the data.

REFERENCES:
- [Background] de Paula LIDS, de Oliveira LF, Cruz BP, de Oliveira DM, Miranda LM, de Moraes Ribeiro M, Duque RO, de Figueiredo AA, de Bessa J Jr, Netto JMB. Parasacral transcutaneous electrical neural stimulation (PTENS) once a week for the treatment of overactive bladder in children: A randomized controlled trial. J Pediatr Urol. 2017 Jun;13(3):263.e1-263.e6. doi: 10.1016/j.jpurol.2016.11.019. Epub 2016 Dec 21. PMID 28089606
- [Background] Farhat W, Bagli DJ, Capolicchio G, O'Reilly S, Merguerian PA, Khoury A, McLorie GA. The dysfunctional voiding scoring system: quantitative standardization of dysfunctional voiding symptoms in children. J Urol. 2000 Sep;164(3 Pt 2):1011-5. doi: 10.1097/00005392-200009020-00023. PMID 10958730

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Urotherapy | Standard Urotherapy + PTENS
Started | 15 | 15
Completed | 11 | 13
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Urotherapy | Standard Urotherapy + PTENS | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 15 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 10 [8.6 to 10.6] | 9.1 [7.6 to 10.6] | 9.55 [8.1 to 10.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 10 | 8 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 13 | 12 | 25
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Initail Dysfunctional Voiding Scoring System Score [Median (Inter-Quartile Range); unit: units on a scale] — Dysfunctional Voiding Symptom Score is a validated clinical questionnaire designed to quantify the severity of pediatric voiding dysfunction on a scale of 0 (non-existent) to 30 (most severe).
  units on a scale | 10 [7.5 to 12.5] | 11 [10 to 13] | 10.5 [8.75 to 12.75]

OUTCOME MEASURES:

1. Primary Outcome: Dysfunctional Voiding Symptom Score
Description: At week 6 a Dysfunctional Voiding Scoring System Score. Descriptive statistics will be used to analyze these data in comparison to pre-study scores.
  As stated above, Dysfunctional Voiding Symptom Score is a validated clinical questionnaire designed to quantify the severity of pediatric voiding dysfunction on a scale of 0 (non-existent) to 30 (most severe).
Time Frame: week 6
Population: Patients who met elegibility criteria and enrolled in the study and then completed the DVSS questionnaire at 6 weeks into the study. These numbers differ from the total number of patients enrolled as there were some who did not complete the 6 week questionnaire.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard Urotherapy | Standard Urotherapy + PTENS
Number analyzed (Participants) | 8 | 7
score on a scale | 8 [5.5 to 11] | 11 [8 to 12]

2. Primary Outcome: Voiding Diary and the Number of Episodes of Incontinence Per Day
Description: 48-hour Voiding Diary and Nighttime Wetting log will be repeated and evaluated. This was added as a separate primary outcome as it is separate from the Dysfunctional Voiding Symptom Score. The voiding diary will be used to evaluate the number of episodes of incontinence per day and descriptive statistics will be used to compare this to pre-study numbers.
Time Frame: week 6, week 12
Population: number of patients who completed 48 hour voiding diary at 6 weeks.
Measure: Median (Inter-Quartile Range); unit: Incontinence Episodes
Arm/Group | Standard Urotherapy | Standard Urotherapy + PTENS
Number analyzed (Participants) | 7 | 11
Incontinence Episodes
  6 week Voiding Diary | 2 [0.5 to 3.5] | 1 [0 to 2]
  12 week Voiding Diary: number analyzed (Participants) | 7 | 10
  12 week Voiding Diary | 1 [0.5 to 2] | 0.5 [0 to 3.75]

3. Secondary Outcome: Secondary Outcome. Review of Adverse Events.
Description: Confirmation of safety and identification of potential adverse events. We will review all data for potential adverse events.
Time Frame: Week 6 through Week 12
Measure: Number; unit: events
Arm/Group | Standard Urotherapy | Standard Urotherapy + PTENS
Number analyzed (Participants) | 11 | 13
events | 0 | 2

ADVERSE EVENTS:
Time Frame: 12 weeks (time that data was collected between enrollment and subjects completing their participation in the study)
Arm/Group | Standard Urotherapy | Standard Urotherapy + PTENS
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/13
Other Adverse Events (participants affected / at risk) | 0/11 | 2/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Urotherapy (N=11) | Standard Urotherapy + PTENS (N=13)
Pruritis at Pad Site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — mild pruritis at pad site (self-limited and not requiring medical intervention)
Discomfort when removing pad (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — mild discomfort from adhesive on skin when removing the TENS pad

LIMITATIONS AND CAVEATS:
Limitations included patients being lost to follow-up or not completing their voiding diaries or DVSS questionnaires so that the number of patients with complete information was only slightly higher than half of the total who were initially enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT04570605/Prot_SAP_001.pdf